CLINICAL TRIAL: NCT00456274
Title: Baselines in Reproductive Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Janet E. Hall, MD, Associate Physician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1999P-003770
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Amenorrhea; Hypogonadotropic Hypogonadism; Kallmann's Syndrome
Keywords: Hypothalamic Amenorrhea; Idiopathic hypogonadotropic hypogonadism; Acquired hypogonadotropic hypogonadism; Kallmann's Syndrome; Amenorrhea; Gonadotropin Releasing Hormone
MeSH Terms: conditions — Amenorrhea; Hypogonadism; Kallmann Syndrome; Idiopathic Hypogonadotropic Hypogonadism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Frequent baseline blood sampling

INTERVENTIONS:
Procedure: Frequent baseline blood sampling — 3 ml of blood sampled every 10 minutes for a total of 8-12 hours

SUMMARY:
The purpose of the study is to explore the way in which gonadotropins (pituitary hormones) are released into the body. The knowledge acquired in this study will be used for the diagnosis and treatment of reproductive endocrine disorders.

We seek to investigate the baseline characteristics of the GnRH-induced gonadotropin pulsations of patients with the following diagnoses:

* Hypothalamic Amenorrhea (HA)
* Idiopathic hypogonadotropic hypogonadism (IHH)
* Polycystic ovarian disease (PCOD)
* Acquired hypogonadotropic hypogonadism (AHH)
* Premature Ovarian Failure (POF)

**WE ARE CURRENTLY RECRUITING ONLY SUBJECTS WITH A DIAGNOSIS OF IHH.**

This has been an extremely productive and pivotal protocol in the studies of female reproductive physiology and pathophysiology and continues to be critical for defining the neuroendocrine abnormalities in patients with reproductive disorders. In some cases, it is also helpful in the planning of subsequent therapy if so desired.

It is important to note that minors have been included in this protocol, as many patients are extremely anxious to know more about their neuroendocrine disorder. With minors who would like to know if their disorder is correctable, this protocol may be followed up with administration of pulsatile gonadotropin-releasing hormone (GnRH).

DETAILED DESCRIPTION:
Normal reproductive cycles in women require the integrated function of the hypothalamus, pituitary and ovaries. The hypothalamic component of the reproductive system can be assessed directly in lower animal species by measurement of gonadotropin releasing hormone (GnRH) directly from pituitary portal blood and recording of multiunit activity from the median eminence of the hypothalamus, providing direct information about the physiology of GnRH secretion and the activity of the GnRH pulse generator. However, these techniques are not feasible in the human. In addition, measurement of GnRH levels in peripheral blood does not accurately reflect hypothalamic GnRH secretion. Thus, indirect methods must be used to gain insight into hypothalamic function in the human.

In the human, pulsatile luteinizing hormone (LH) secretion has been used as a mirror of hypothalamic GnRH secretion, citing comparative data from the rat, sheep, and non-human primate which indicate that pulses of LH are directly linked to antecedent pulses of GnRH. LH secretion thus provides an estimate of the underlying frequency of GnRH pulse generator activity provided that the assay is sufficiently precise, with a low coefficient of variation, and that blood sampling is frequent enough to accurately reflect the underlying frequency of episodic GnRH pulsatility. The use of pulsatile secretion of the free alpha subunit (FAS) of the gonadotropins has recently been proposed as an alternative and improved marker of GnRH secretion in the human due to a half-life of 15 minutes versus 20 to 40 minutes for LH. Despite the dual control of FAS by GnRH and thyroid releasing hormone (TRH), our studies have shown that the pulsatile component of FAS secretion is driven solely by GnRH in euthyroid subjects. Such studies have indicated:

1. the nearly complete concordance of pulses of FAS with those of LH in normal women, and in GnRH-deficient subjects undergoing GnRH replacement;
2. the absence of pulsatile secretion of FAS in GnRH-deficient subjects; and
3. the abolition of pulsatile FAS secretion in concert with that of LH following administration of a GnRH antagonist in normal and postmenopausal women.

We have proposed that abnormalities in the pulsatile secretion of GnRH underlie many reproductive abnormalities and that these may explain the clinical variability, which exists even within a given diagnostic category. In this protocol, we have sought to define the specific neuroendocrine profile in patients with amenorrhea or oligomenorrhea. In some patients, the results of these studies can then correlated with clinical outcomes of ovulation induction protocols and with genotype information. We have examined the spectrum of abnormal patterns of LH (and by inference GnRH) secretion in women with secondary hypogonadotropic hypogonadism. In 73 studies in 50 women, it has been determined that the most common neurosecretory defect is low frequency/low amplitude followed by normal frequency/normal amplitude, apulsatile, and low amplitude/normal frequency. Of patients studied on several occasions, 75% demonstrated at least 2 different patterns of LH secretion and 33% reverted at least once to a normal pattern of secretion. Study of the baseline patterns of LH secretion in patients with acquired GnRH deficiency/acquired hypothalamic hypogonadism (AHH) indicates that this group of patients has either an apulsatile pattern or a pattern of low amplitude LH pulses in comparison with normal women in the early follicular phase (matched for ovarian steroid levels). In these patients, the specific LH pattern does not predict response to pulsatile GnRH used for ovulation induction. FAS is apulsatile in the majority of patients with primary amenorrhea and absent LH pulses providing further support for the hypothesis that the pulsatile component of FAS secretion is primarily driven by GnRH in euthyroid patients despite the dual control of FAS by GnRH and TRH. As in men with presumed GnRH deficiency, occasional patients with absent LH pulses will have FAS pulses. These interesting patients are being further evaluated with respect to their pattern of TSH secretion and the bioactivity of their LH.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women between the ages of 16-45 years
* Negative pregnancy test
* On no gonadal steroid preparations for at least 3 months, with the exception of the idiopathic hypogonadotropic hypogonadism (IHH) group, they should be off gonadal steroid for at least 4 weeks

The following test will be performed if they had not been done in the last 2 months

* Normal blood count
* Normal thyroid function test

Exclusion Criteria:

* Hemoglobin levels less than 11 gm/dL
* Positive pregnancy test
* Abnormal thyroid function
* Abnormal MRI (IHH)

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 1999-09; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Number of luteinizing hormone (LH) and FAS (free alpha subunit) pulses | 8-12 hours

SECONDARY OUTCOMES:
Amplitude of LH and FAS pulses | 8-12 hours
Inter-pulse interval for LH and FAS pulses | 8-12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Hall, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Clarke IJ. Variable patterns of gonadotropin-releasing hormone secretion during the estrogen-induced luteinizing hormone surge in ovariectomized ewes. Endocrinology. 1993 Oct;133(4):1624-32. doi: 10.1210/endo.133.4.8404603.
- [Background] Wilson RC, Kesner JS, Kaufman JM, Uemura T, Akema T, Knobil E. Central electrophysiologic correlates of pulsatile luteinizing hormone secretion in the rhesus monkey. Neuroendocrinology. 1984 Sep;39(3):256-60. doi: 10.1159/000123988. PMID 6504270
- [Background] Nett TM, Adams TE. Further studies on the radioimmunoassay of gonadotropin-releasing hormone: effect of radioiodination, antiserum and unextracted serum on levels of immunoreactivity in serum. Endocrinology. 1977 Oct;101(4):1135-44. doi: 10.1210/endo-101-4-1135. No abstract available. PMID 332491
- [Background] Adams JM, Taylor AE, Schoenfeld DA, Crowley WF Jr, Hall JE. The midcycle gonadotropin surge in normal women occurs in the face of an unchanging gonadotropin-releasing hormone pulse frequency. J Clin Endocrinol Metab. 1994 Sep;79(3):858-64. doi: 10.1210/jcem.79.3.7521353.
- [Background] Filicori M, Flamigni C, Crowley WF, Jr. The critical role of blood sampling frequency in the estimation of episodic luteinizing hormone secretion in normal women. In: Crowley Jr WF, Hofler JG (eds) The Episodic Secretion of Hormones. New York: Churchill Livingston.5-13, 1987.
- [Background] Hall JE, Lavoie HB, Marsh EE, Martin KA. Decrease in gonadotropin-releasing hormone (GnRH) pulse frequency with aging in postmenopausal women. J Clin Endocrinol Metab. 2000 May;85(5):1794-800. doi: 10.1210/jcem.85.5.6612. PMID 10843154
- [Background] Whitcomb RW, O'Dea LS, Finkelstein JS, Heavern DM, Crowley WF Jr. Utility of free alpha-subunit as an alternative neuroendocrine marker of gonadotropin-releasing hormone (GnRH) stimulation of the gonadotroph in the human: evidence from normal and GnRH-deficient men. J Clin Endocrinol Metab. 1990 Jun;70(6):1654-61. doi: 10.1210/jcem-70-6-1654. PMID 1693373
- [Background] Crowley WF, Taylor AE, Martin KA, Whitcomb RW, Finkelstein JS, Hall JE. 1994 Use of the free alpha subunit (FAS) of glycoprotein secreting hormones as a surrogate marker of GnRH secretion in the human. In: Glycoprotein Hormones: Structure, Function and Clinical Implications. JW Lusbader, LD Puett, R Ruddon (eds), Serono Symposia, UAS pp. 253-63.
- [Background] Sharpless JL, Supko JG, Martin KA, Hall JE. Disappearance of endogenous luteinizing hormone is prolonged in postmenopausal women. J Clin Endocrinol Metab. 1999 Feb;84(2):688-94. doi: 10.1210/jcem.84.2.5433. PMID 10022439
- [Background] Kourides IA, Weintraub BD, Re RN, Ridgway EC, Maloof F. Thyroid hormone, oestrogen, and glucocorticoid effects on two different pituitary glycoprotein hormone alpha subunit pools. Clin Endocrinol (Oxf). 1978 Dec;9(6):535-42. doi: 10.1111/j.1365-2265.1978.tb01511.x. No abstract available. PMID 747894
- [Background] Hall JE, Whitcomb RW, Rivier JE, Vale WW, Crowley WF Jr. Differential regulation of luteinizing hormone, follicle-stimulating hormone, and free alpha-subunit secretion from the gonadotrope by gonadotropin-releasing hormone (GnRH): evidence from the use of two GnRH antagonists. J Clin Endocrinol Metab. 1990 Feb;70(2):328-35. doi: 10.1210/jcem-70-2-328. PMID 2105329
- [Background] Hall JE, Martin KA, Whitney HA, Landy H, Crowley WF Jr. Potential for fertility with replacement of hypothalamic gonadotropin-releasing hormone in long term female survivors of cranial tumors. J Clin Endocrinol Metab. 1994 Oct;79(4):1166-72. doi: 10.1210/jcem.79.4.7962290.
- [Background] Perkins RB, Hall JE, Martin KA. Neuroendocrine abnormalities in hypothalamic amenorrhea: spectrum, stability, and response to neurotransmitter modulation. J Clin Endocrinol Metab. 1999 Jun;84(6):1905-11. doi: 10.1210/jcem.84.6.5823. PMID 10372685
- [Background] Hayes FJ, McNicholl DJ, Schoenfeld D, Marsh EE, Hall JE. Free alpha-subunit is superior to luteinizing hormone as a marker of gonadotropin-releasing hormone despite desensitization at fast pulse frequencies. J Clin Endocrinol Metab. 1999 Mar;84(3):1028-36. doi: 10.1210/jcem.84.3.5579. PMID 10084591
- See also: MGH Reproductive Endocrine Research Studies — http://www.massgeneral.org/reproendo/pages/reu_study_subject.htm